CLINICAL TRIAL: NCT02423265
Title: The Effectiveness of Ranolazine in Reducing Cardiac Ischaemia Induced by Chronic Total Occlusions of Coronary Arteries
Brief Title: Efficacy of Ranolazine in Patients With Chronic Total Occlusions of Coronary Arteries
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: slow recruitment; local new issues with CMR after study start
Sponsor: East Carolina University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Dr Ashesh N. Buch, Assistant Professor Cardiovascular Sciences (Interventional Cardiology), East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IN-US-259-0172 Buch ISR; UMCIRB 13-001574 (Other: Institutional Review Board (IRB))
Record Dates: First submitted 2015-04-12; First posted 2015-04-22 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Myocardial Ischemia; Coronary Artery Disease; Arteriosclerosis; Chronic Stable Angina
Keywords: Chronic total coronary occlusions; Ranolazine
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Arteriosclerosis; Angina, Stable | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Active Comparator): 500mg bd ranolazine for 1 week then uptitrated to 1000mg bd to continue for 8 weeks
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Matching placebo, with up titration after 1 week as in active treatment arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ranolazine — Ranolazine: 500 mg twice day, up-titrated after 1 week to 1000 mg twice a day
  Other Names: Renexa
  Arms: Ranolazine
Drug: Placebo — Matching placebo: up-titration after 1 week
  Arms: Placebo

SUMMARY:
Anti-anginal drugs relieve ischemia and symptoms by reducing myocardial oxygen demand by reducing heart rate and or contractility (beta-blockers, phenylalkylamine and benzothiazepineate classes of calcium antagonists) or vasodilatation of the venous system (fall in pre-load) and coronary vessels.

Late sodium channels remain open for longer in the presence of myocardial ischaemia. Ranolazine, a novel anti-anginal agent, acts by inhibiting the inward late inward sodium current (INaL), reducing intracellular sodium accumulation and consequently intracellular calcium overload via the sodium/calcium exchanger. It is currently thought that this reduction in intracellular calcium reduces diastolic myocardial stiffness and therefore compression of the small coronary vessels. There is considerable animal data to support this theory.

There are good theoretical reasons to postulate that patients with chronically occluded vessels may derive less benefit from conventional anti-anginal agents, particularly vasodilators. The ischemic myocardium, subtended by the occluded vessel, will already be subject to significant concentrations of paracrine vasodilators such as adenosine. Ranolazine, therefore, may on the basis of its mechanism of action, provide greater relief of ischemia in such patients than conventional anti-anginal agents.

DETAILED DESCRIPTION:
To test this hypothesis, a randomized study comparing addition of ranolazine to addition of a minimum of 2 conventional anti-anginal agents in patients with chronic total occlusions would be required. To be sufficiently powered, this would require a significant number of patients recruited in a multi-center trial. This study is an initial pilot study with inactive placebo, not addition of a conventional anti-anginal agent, as the control using MRI imaging data as the primary end-point.

ELIGIBILITY:
Inclusion Criteria:

* Angiographically proven coronary artery disease with chronic stable angina for at least 3 months.
* Abnormal stress test (treadmill ECG, nuclear stress test, dobutamine stress echocardiogram or stress perfusion cardiac MRI)
* ≥ 1 chronically occluded coronary artery of a dominant coronary vessel or the left anterior descending artery and/or ≥ 1 occluded vein graft to chronically occluded native coronary vessel
* Subjects must be taking a minimum of 2 anti-anginal agents:

Exclusion Criteria:• Coronary revascularization in the preceding 2 months

* LVEF < 40
* Terminal illness such as cancer
* Occluded recessive coronary vessel
* Hepatic insufficiency,
* Liver cirrhosis,
* Prolonged QT interval on ECG,
* Severe renal failure (see below), Excluding patients with CrCl < 30
* Drugs that are strong inhibitors of CYP3A such as, ketoconazole, macrolide antibiotics and HIV protease inhibitors.
* Limit Ranolazine to 500mg BID in patients on concurrent diltiazem/verapamil
* Limit concurrent simvastatin to 20 mg/day
* Limit concurrent metformin to 1700 mg/day
* Inability to have an MRI scan/known claustrophobia

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Cardiac MRI (CMR) strain | 8 weeks
  The extent of reversibly ischaemic LV myocardium will be assessed using CMR strain at rest and stress

SECONDARY OUTCOMES:
Dobutamine wall motion scoring index (WMSI) | 8 weeks
  CMR derived end point
Quality of Life/burden of angina | 8 weeks
  QoL questionnaire based assessment (Seattle Angina Quesstionnaire, SAQ; Duke Activity Status Index, DASI;Medical Outcomes Study-Short Form12 )
Treadmill ECG exercise distance | 8 weeks
  Functional capacity assessment
Time to ECG changes (ST depression) on exercise ECG | 8 weeks
  If baseline ECG permits, this will allow assessment of impact of treatment on ECG markers of ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Ashesh N Buch, MB.ChB, M.D., Principal Investigator — East Carolina University
Locations (1):
- East Carolina Heart Institute at Vidant Medical Center, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided